CLINICAL TRIAL: NCT06369168
Title: Effect and Effectiveness of Auricular Acupuncture in Improving Hot Flashes During Adjuvant Endocrine Therapy in Women With Breast Cancer: A Randomized Controlled Study
Brief Title: Auricular Acupuncture and Hot Flashes During Adjuvant Endocrine Therapy
Acronym: OhrHit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kliniken Essen-Mitte
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Hot Flashes
Keywords: breast cancer; hot flashes; acupuncture; endocrine therapy
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms | interventions — Acupuncture, Ear

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NADA auricular acupuncture (Active Comparator): Patients in one intervention group are treated twice a week for five weeks with balanced ear acupuncture.The data sets of those subjects who received at least eight balanced ear acupuncture treatments will be compared with those who got NADA acupuncture and those who were not treated.
  Interventions: Device: auricular acupuncture
- balanced auricular acupuncture (Active Comparator): Patients in the other intervention group are treated twice a week for five weeks with NADA ear acupuncture. The data sets of those subjects who received at least eight NADA ear acupuncture treatments will be compared with those who got balanced ear acupuncture and those who were not treated.
  Interventions: Device: auricular acupuncture
- wait list control (No Intervention): Control group: At the end of the 3-month follow-up, the patients in the control group received 10 ear acupuncture treatments in a group setting.

INTERVENTIONS:
Device: auricular acupuncture — two auricular acupuncture methods are compared with each other and with no treatment
  Arms: NADA auricular acupuncture; balanced auricular acupuncture

SUMMARY:
With this clinical trial we investigate whether auricular acupuncture during adjuvant endocrine therapy has an improving effect on hot flashes, which are often perceived as psychologically and physically stressful in self-assessment of women with breast cancer.

Empirical studies indicate that body acupuncture has positive effects on hot flashes. As auricular acupuncture offers a number of advantages over body acupuncture, a three-armed randomised controlled research design is being used to investigate whether hot flashes caused by endocrine therapy are also reduced by ear acupuncture. Balanced ear acupuncture will be compared with NADA ear acupuncture in terms of efficacy and effectiveness. In addition, the effects of the two forms of therapy on the patients' individual quality of life, fatigue, stress perception and sleep quality will be analysed.

DETAILED DESCRIPTION:
In Germany, one in eight women will develop breast cancer in her lifetime, with a relative 5-year survival rate of 88%. Around 70 % of breast cancer cases are hormone receptor positive. Adjuvant endocrine therapy is recommended to reduce the risk of recurrence.The results of a systematic review show that around 52.4 % to 84.8 % of patients adhere to the treatment. It was also shown that non-adherence to treatment has a negative impact on the risk of breast cancer recurrence and the development of distant metastases, as well as on mortality. Lack of adherence to treatment is related, among other things, to the side effects of endocrine therapy, which significantly reduce quality of life. In particular, musculoskeletal syndrome and sleep disorders lead to discontinuation of endocrine treatment with an aromatase inhibitor. Many patients also suffer from hot flashes, sexual dysfunction, weight gain, bone density loss, depression, cognitive dysfunction and fatigue.

The study focuses on hot flashes, which have a negative impact on sleep and promote symptoms of fatigue. Due to the endocrine therapy, the symptoms are usually more pronounced than the menopause-related symptoms. However, oestrogen-based hormone replacement therapy is contraindicated, while non-hormonal medication such as venlafaxine or gabapentin often have serious side effects. An alternative is body acupuncture, which can decrease hot flashes in women with breast cancer. One of the advantages of acupuncture compared to drug treatments is that it is considered having very few side effects.

With the help of a three-armed randomized controlled research design, this study aims to investigate the efficacy and effectiveness of balanced ear acupuncture compared to NADA ear acupuncture in the treatment of hot flashes caused by endocrine therapy. In addition, the effects of the two forms of therapy on the individual quality of life, fatigue, stress perception and sleep quality of the patients will be analyzed.The respective results will be compared with those of a control group that did not receive acupuncture during the observation period.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of non-metastatic hormone receptor-positive breast CA (TNM stage I-III) under adjuvant endocrine therapy
* hot flashes, measured with the MRS (Menopause Rating Scale)
* willingness to participate in the study and signed informed consent

Exclusion Criteria:

* ongoing or planned chemotherapy, radiotherapy, follow-up treatment or reconstructive plastic surgery during the study period
* severe physical or psychopharmacologically treated psychiatric comorbidity, due to which a patient is unable to participate in the study
* pregnancy
* participation in other clinical trials with behavioural, psychological or complementary medicine, psychological or complementary medical interventions
* regular use of barbiturates, antidepressants, abuse of drugs and/or alcohol
* ongoing acupuncture treatment
* lack of ability to complete the questionnaires independently
* operations or infections in the area to be acupunctured

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 107 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
subscale somato-vegetative symptoms of the Menopause Rating Scale (MRS) | Baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  measure for hot flashes, from minimum 0 to maximum 4, with the maximum being the worst outcome

SECONDARY OUTCOMES:
Menopause Rating Scale (MRS) total score | Baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  self-administered scale to assess menopausal symptoms and complaints, to evaluate the severity of symptoms over time, and to measure changes pre- and postmenopause replacement therapy, from minimum 0 to maximum 4 with the maximum being the worst outcome
Psychological symptoms and urogenital symptoms subscales of the MRS | Baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  subscale of the MRS, from minimum 0 to maximum 4, with the maximum being the worst outcome
functional assessment of cancer therapy - breast (FACT-B) | Baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  Quality of life; physical and emotional wellbeing: from minimum 0 to maximum 4, with the maximum being the worst outcome, social relationships, sexual life satisfaction, and functionality: from minimum 0 to maximum 4, with the maximum being the best outcome
perceived stress questionnaire (PSQ) | Baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  stress, from minimum 0 to maximum 4, with the maximum being the strongest agreement to the statements
insomnia severity index (ISI) | Baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  insomnia severity, from minimum 0 to maximum 4, with the maximum being the worst outcome
big five inventory (BFI) | current condition at baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  fatigue, with minimum 1 to maximum 10, with the maximum being the worst outcome
Expected effect of the respective intervention on a 100mm visual analogue scale | baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  expected effect of the treatment and fulfilling of the expectation, from minimum 1 to maximum 10, with the maximum being the highest expectation
intensity and degree of impairment due to hot flashes on a 100mm visual analogue scale | current condition at baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  individual extent of hot flashes, from minimum 1 to maximum 10, with the maximum being the worst outcome
adverse events (AEs) | current condition at baseline, end of the intervention (6 weeks after the beginning), three months follow-up
  negative side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Evang. Kliniken Essen-Mitte gGmbH, Essen, Germany